CLINICAL TRIAL: NCT03173664
Title: Post-Approval Study of Clinical Outcomes and Visual Symptoms With the KAMRA Inlay
Brief Title: Post-Approval Study With the KAMRA Inlay
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: AcuFocus, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: KAMR-203-PASQ
Record Dates: First submitted 2017-05-25; First posted 2017-06-02 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: KAMRA Inlay — Unilateral implantation of the KAMRA inlay in the corneal stroma.

SUMMARY:
KAMRA inlay, to be unilaterally implanted into the cornea of a subject's non-dominant eye. The inlay is to be inserted into a stromal pocket created with a surgical femtosecond laser.

DETAILED DESCRIPTION:
This is a post-approval study of the KAMRA inlay performance and potential device-related issues in a broader population over an extended period of time after pre-market establishment of reasonable safety and effectiveness.

Study objectives include:

* Evaluate the long-term performance (effectiveness) and safety of the device;
* Evaluate real-world performance of the device in subjects treated by refractive surgeons with a range of experience levels;
* Evaluate the performance of the device in racial/ethnic subgroups representative of the population for which the device is intended.

In addition, the data from a subset of the first 105 subjects who have been enrolled in this study will be used to validate the KAMRA Inlay Patient Questionnaire (KIPQ) for the assessment of patients who have received the KAMRA inlay for the treatment of presbyopia.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the indications for use for this device;
2. Do not have any of the conditions described in the contraindications in the labeling of the device;
3. Are willing and able to provide informed consent;
4. Are not participating in any other clinical studies during the course of the study.

Exclusion Criteria:

1. Subject has insufficient ability to read or write that would prevent them from completing a questionnaire without help; or
2. Subject is not a fluent speaker of U.S. English.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Phakic, presbyopic patients between the ages of 45 and 60 years old who have cycloplegic refractive spherical equivalent of +0.50 diopters to -0.75 diopters with less than or equal to 0.75 diopters of refractive cylinder, who do not require glasses or contact lenses for clear distance vision, and who require near correction of +1.00 to +2.50 diopters of reading add.
Sampling Method: Probability Sample
Enrollment: 529 (Estimated)
Dates: Start 2018-07-31 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Monocular Near Visual Acuity | Five years
  Percentage of implanted eyes with monocular near visual acuity of 20/40 or better is greater than or equal to 75% of implanted eyes.

SECONDARY OUTCOMES:
Best-corrected distance visual acuity | Five years
  Percentage of implanted eyes with a persistent loss of two or more lines of best-corrected distance visual acuity from baseline at the subject's last study visit is less than 5%.

CONTACTS AND LOCATIONS:
Overall Officials: TBD TBD, M.D., Principal Investigator

IPD SHARING:
Plan to Share IPD: No